CLINICAL TRIAL: NCT01059955
Title: Iontophoresis Delivery of Dexamethasone Phosphate for Non-infectious, Non-necrotizing Anterior Scleritis, Phase 1 Dose-varying Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Kempen (Other)
Responsible Party: Sponsor-Investigator, John Kempen, Associate Professor of Ophthalmology and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-IST-001; 1R01FD003910 (FDA)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Non-infectious, Non-necrotizing Anterior Scleritis
Keywords: scleritis; anterior scleritis; nodular anterior scleritis; diffuse anterior scleritis
MeSH Terms: conditions — Scleritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment at day 0 and day 7 (Experimental): Iontophoresis Delivery of Dexamethasone Phosphate (EGP-437) at one of three different iontophoretic doses. One treatment will be given at Day 0 (baseline) and one at Day 7.
  The three iontophoresis doses are:
  1. Ocular iontophoresis with EGP-437 1.2 mA-min at 0.4 mA
  2. Ocular iontophoresis with EGP-437 2.5 mA-min at 0.8 mA
  3. Ocular iontophoresis with EGP-437 4.5 mA-min at 1.5 mA
  Interventions: Drug: Dexamethasone Phosphate Ophthalmic Solution (EGP-437)
- Active Treatment at Day 0, Sham Treatment at Day 7 (Active Comparator): Iontophoresis Delivery of Dexamethasone Phosphate (EGP-437) at one of three different iontophoretic doses. One treatment will be given at Day 0 (baseline) and a sham treatment Day 7.
  The three iontophoresis doses are:
  1. Ocular iontophoresis with EGP-437 1.2 mA-min at 0.4 mA
  2. Ocular iontophoresis with EGP-437 2.5 mA-min at 0.8 mA
  3. Ocular iontophoresis with EGP-437 4.5 mA-min at 1.5 mA
  Interventions: Drug: Dexamethasone phosphate ophthalmic solution

INTERVENTIONS:
Drug: Dexamethasone Phosphate Ophthalmic Solution (EGP-437) — Transcleral iontophoretic delivery of dexamethasone phosphate ophthalmic solution. Dexamethasone phosphate ophthalmic solution as a ready to use 40 mg/mL solution (preservative free and intended for single-use only).
  Arms: Active treatment at day 0 and day 7
Drug: Dexamethasone phosphate ophthalmic solution — Transcleral iontophoretic delivery of dexamethasone phosphate ophthalmic solution. Dexamethasone phosphate ophthalmic solution as a ready to use 40 mg/mL solution (preservative free and intended for single-use only)
  Arms: Active Treatment at Day 0, Sham Treatment at Day 7

SUMMARY:
This is an initial clinical trial evaluating whether different doses of iontophoresis for delivery of dexamethasone phosphate can be tolerated by eyes of patients with non-infections, non-necrotizing scleritis. A secondary goal is to get preliminary information about whether the treatment is likely to be an effective treatment for scleritis. If the results are favorable, further trials evaluating the treatment may be pursued.

Funding sources: FDA OOPD, Eyegate Pharmaceuticals, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age at least 18 years
2. A diagnosis of active non-infectious, non-necrotizing anterior scleritis (nodular or diffuse is acceptable)
3. Not planning to undergo elective ocular surgery during the study
4. Provide written informed consent
5. Be able and willing to follow instructions, return for all study visits, and willing to comply with all study-related instructions
6. If female and of childbearing potential; submit a urine sample and have a negative pregnancy test at Visit 1; agree to use an acceptable method of contraception during the study. A woman is considered of childbearing potential unless she is surgically sterile (hysterectomy or tubal ligation) or is post-menopausal (has not had a menstrual cycle for >2 years or has laboratory evidence of a post-menopausal state). Acceptable methods of contraception include: spermicide with barrier, hormonal contraception, IUD, or surgical sterilization of partner. Complete abstinence throughout the study period also is acceptable.

Exclusion Criteria:

1. Contraindications to the use of the test articles
2. Known allergy or sensitivity to any medication used in this study, including the study medication or its components (e.g., corticosteroids)
3. For patients not taking systemic corticosteroids or immunosuppressants, any condition constituting conferring a likelihood that systemic corticosteroids or immunosuppressants would need to be started during the 56-day study period
4. For patients already taking systemic corticosteroids and/or immunosuppressants, any condition conferring a likelihood that systemic corticosteroid or immunosuppressant dosage would need to be changed during the 56-day study period
5. Intraocular pressure high enough that intraocular pressure-lowering medications are likely to be needed (≥25 mmHg or IOP>target pressure for patients with glaucoma); and/or more than two ocular anti-hypertensive medications (prior IOP-lowering surgery is acceptable; combinations of two agents such as Cosopt or Combigan are considered two medications)
6. Glaucoma sufficiently advanced that an intraocular pressure spike would potentially put the patient at substantial risk of vision loss, per the clinician-investigator's judgment.
7. Cancer
8. Subject is planning to undergo elective surgery during the study period
9. Any active ocular infections (bacterial, viral, or fungal), active ocular inflammation other than scleritis (i.e., follicular conjunctivitis, iritis), or preauricular lymphadenopathy
10. History or diagnosis of ocular herpes or corneal lesion of suspected herpetic origin
11. Severe eyelid or ocular surface lesions impeding application of the iontophoresis applicator
12. Severe / serious ocular pathology or medical condition which may preclude study completion
13. Any condition conferring a likelihood that topical ophthalmic medications in use at baseline would need to be changed during the 56-day study period.
14. History of Stevens-Johnson Syndrome or mucous membrane pemphigoid
15. Unwilling to discontinue use of contact lenses for the duration of the study
16. Any open wounds / skin disease on the forehead where the iontophoresis return electrode will be applied
17. Pacemakers and/or any other electrical sensitive support system
18. Any significant illness or condition that could, in the investigator's or sub-investigator's opinion, be expected to interfere with the study parameters or study conduct; or put the subject at significant risk
19. Be currently pregnant, nursing, or planning a pregnancy; or woman who has a positive pregnancy test
20. Participation in an investigational drug or device study within 30 days of entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 56 days

SECONDARY OUTCOMES:
Improvement on scleritis scale score | 56 days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Wilmer Eye Institute/Johns Hopkins University, Baltimore, Maryland
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health & Sciences University, Portland, Oregon
  - Scheie Eye Institute/University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] O'Neil EC, Huang J, Suhler EB, Dunn JP Jr, Perez VL, Gritz DC, McWilliams K, Peskin E, Ying GS, Bunya VY, Maguire MG, Kempen JH. Iontophoretic delivery of dexamethasone phosphate for non-infectious, non-necrotising anterior scleritis, dose-finding clinical trial. Br J Ophthalmol. 2018 Aug;102(8):1011-1013. doi: 10.1136/bjophthalmol-2017-311610. Epub 2018 Apr 17. PMID 29666122